CLINICAL TRIAL: NCT01061723
Title: A Randomized Double Blind-placebo Controlled Dose Ranging Study to Evaluate the Efficacy and Safety of SAR153191 in Participants With Ankylosing Spondylitis (AS)
Brief Title: Dose Ranging Study to Evaluate the Efficacy and Safety of SAR153191 (REGN88) in Patients With Ankylosing Spondylitis
Acronym: ALIGN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRI11073; 2009-016068-35 (EudraCT Number)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo (for sarilumab) weekly (qw) for 12 weeks.
  Interventions: Drug: Placebo
- Sarilumab 100 mg q2w (Experimental): Sarilumab 100 mg Subcutaneous (SC) injection alternating with placebo every other week (q2w) for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 150 mg q2w (Experimental): Sarilumab 150 mg SC injection alternating with placebo q2w for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 100 mg qw (Experimental): Sarilumab 100 mg SC injection qw for 12 weeks.
  Interventions: Drug: Sarilumab
- Sarilumab 200 mg q2w (Experimental): Sarilumab 200 mg SC injection alternating with placebo q2w for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo
- Sarilumab 150 mg qw (Experimental): Sarilumab 150 mg SC injection qw for 12 weeks.
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Other Names: SAR153191; REGN88
  Arms: Sarilumab 100 mg q2w; Sarilumab 100 mg qw; Sarilumab 150 mg q2w; Sarilumab 150 mg qw; Sarilumab 200 mg q2w
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Subcutaneous
  Arms: Placebo; Sarilumab 100 mg q2w; Sarilumab 150 mg q2w; Sarilumab 200 mg q2w

SUMMARY:
Primary objective:

- to evaluate the efficacy of Sarilumab in participants with Ankylosing Spondylitis (AS) using the assessment in AS working group criteria (ASAS) 20% response criteria (ASAS20)

Secondary objectives:

* to demonstrate that Sarilumab was effective on:

  * assessment of higher level of response [ASAS 40% response criteria (ASAS40)]
  * partial remission
  * disease activity
  * range of motion
  * Magnetic Resonance Imaging (MRI) of the spine
* to assess the safety and tolerability of Sarilumab in participants with AS as well as the pharmacokinetic profile of Sarilumab in participants with AS

DETAILED DESCRIPTION:
The duration of participation in this study for each participant was approximately 22 weeks; including up to 4 weeks screening period, 12-weeks double-blind treatment period and 6-weeks safety follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of AS according to the New York modified criteria
* Participants must had an adequate trial of at least 2 different Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) taken for at least 2 weeks in each case and, on a stable dose for ≥2 weeks or be intolerant to NSAIDs
* Participants must had active AS for ≥3 months before screening and active disease must be present at screening and at baseline; Active AS being defined by:

  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of ≥4 (Numerical Rating Scale 0-10)
  * Total back pain score ≥4 (Numerical Rating Scale 0-10)

Participants treated with corticosteroid must be on a stable dose for ≥2 weeks prior to baseline

Participants treated with the Disease Modifying Anti-Rheumatic Drugs (DMARDs) hydroxychloroquine, sulfasalazine and methotrexate (MTX) must be on stable dose ≥12 weeks prior to baseline

Exclusion criteria:

* <18 years old or ≥75 years old
* Complete fusion of the spine
* Past history of non response to any anti-Tumor Necrosis Factors (TNFs) treatment or non response to any other biological treatment for AS
* Any past or current treatment with anti-TNF's or any biological agent within 3 months prior to screening
* Treatment with DMARDs except for hydroxychloroquine, sulfasalazine and MTX
* MTX >25 mg/week
* hydroxychloroquine >400 mg/day
* Sulfasalazine >3 g/day
* Treatment with oral prednisone or equivalent corticosteroids >10 mg/day within 6 weeks prior to screening
* Use of intramuscular or intra-articular corticosteroids within the last 4 weeks before screening
* Previous treatment with cyclosporine, azathioprine

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (80):
- United States (26):
  - Investigational Site Number 840006, Birmingham, Alabama
  - Investigational Site Number 840033, Anaheim, California
  - Investigational Site Number 840027, Los Angeles, California
  - Investigational Site Number 840007, San Diego, California
  - Investigational Site Number 840013, San Francisco, California
  - Investigational Site Number 840017, Upland, California
  - Investigational Site Number 840009, Boca Raton, Florida
  - Investigational Site Number 840001, Naples, Florida
  - Investigational Site Number 840032, Orlando, Florida
  - Investigational Site Number 840015, Boise, Idaho
  - Investigational Site Number 840021, Rock Island, Illinois
  - Investigational Site Number 840018, Kansas City, Kansas
  - Investigational Site Number 840003, Wheaton, Maryland
  - Investigational Site Number 840029, Worcester, Massachusetts
  - Investigational Site Number 840008, Lansing, Michigan
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840028, Freehold, New Jersey
  - Investigational Site Number 840016, Albany, New York
  - Investigational Site Number 840036, Syracuse, New York
  - Investigational Site Number 840010, Toledo, Ohio
  - Investigational Site Number 840005, Oklahoma City, Oklahoma
  - Investigational Site Number 840023, Bethlehem, Pennsylvania
  - Investigational Site Number 840014, Duncansville, Pennsylvania
  - Investigational Site Number 840004, Dallas, Texas
  - Investigational Site Number 840030, Houston, Texas
  - Investigational Site Number 840034, Chesapeake, Virginia
- Australia (4):
  - Investigational Site Number 036003, Hobart
  - Investigational Site Number 036001, Malvern East
  - Investigational Site Number 036004, Shenton Park
  - Investigational Site Number 036002, Woolloongabba
- Austria (2):
  - Investigational Site Number 040001, Graz
  - Investigational Site Number 040002, Vienna
- Belgium (5):
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056005, Genk
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056002, Leuven
  - Investigational Site Number 056004, Liège
- Canada (10):
  - Investigational Site Number 124007, London
  - Investigational Site Number 124004, Montreal
  - Investigational Site Number 124008, Newmarket
  - Investigational Site Number 124003, Pointe-Claire
  - Investigational Site Number 124001, Québec
  - Investigational Site Number 124006, Saskatoon
  - Investigational Site Number 124005, Toronto
  - Investigational Site Number 124009, Trois-Rivières
  - Investigational Site Number 124002, Vancouver
  - Investigational Site Number 124010, Vancouver
- Czechia (5):
  - Investigational Site Number 203003, Brno
  - Investigational Site Number 203005, Hlučín
  - Investigational Site Number 203002, Hradec Králové
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203004, Uherské Hradiště
- France (4):
  - Investigational Site Number 250001, Besançon
  - Investigational Site Number 250005, Bordeaux
  - Investigational Site Number 250002, Créteil
  - Investigational Site Number 250003, Paris
- Germany (5):
  - Investigational Site Number 276002, Berlin
  - Investigational Site Number 276004, Erlangen
  - Investigational Site Number 276003, Frankfurt am Main
  - Investigational Site Number 276005, Hamburg
  - Investigational Site Number 276001, Herne
- Hungary (4):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348003, Debrecen
  - Investigational Site Number 348005, Sátoraljaújhely
  - Investigational Site Number 348004, Veszprém
- Lithuania (2):
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440002, Vilnius
- Netherlands (2):
  - Investigational Site Number 528001, Amsterdam
  - Investigational Site Number 528002, Nijmegen
- Poland (5):
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616001, Krakow
  - Investigational Site Number 616004, Lublin
  - Investigational Site Number 616005, Torun
  - Investigational Site Number 616003, Warsaw
- Spain (4):
  - Investigational Site Number 724004, A Coruña
  - Investigational Site Number 724005, Barcelona
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724001, Seville
- Turkey (Türkiye) (2):
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792001, Izmir

REFERENCES:
- [Result] Sieper J, Braun J, Kay J, Badalamenti S, Radin AR, Jiao L, Fiore S, Momtahen T, Yancopoulos GD, Stahl N, Inman RD. Sarilumab for the treatment of ankylosing spondylitis: results of a Phase II, randomised, double-blind, placebo-controlled study (ALIGN). Ann Rheum Dis. 2015 Jun;74(6):1051-7. doi: 10.1136/annrheumdis-2013-204963. Epub 2014 Feb 18. PMID 24550171

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 68 centers in Europe, Canada and the United States. A total of 563 participants were screened between 04 February 2010 and 24 February 2011. Of 563 participants, 301 were randomized and 300 were treated.
Pre-assignment Details: Participants were randomized in 1:1:1:1:1:1 ratio for Placebo and Sarilumab (100 mg weekly [qw]; 150 mg qw; 100 mg every other week [q2w]; 150 mg q2w and 200 mg q2w) with screening high-sensitivity C-Reactive Protein (hs-CRP) (≤1.5 mg/L or >1.5 mg/L) and region as stratification factors.
Groups:
- Placebo: Placebo (for sarilumab) qw for 12 weeks.
- Sarilumab 100 mg q2w: Sarilumab 100 mg subcutaneous (SC) injection alternating with placebo q2w for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Started | 50 | 49 | 50 | 52 | 50 | 50
Treated | 50 | 49 | 50 | 52 | 50 | 49
Completed | 46 | 43 | 40 | 44 | 47 | 41
Not Completed | 4 | 6 | 10 | 8 | 3 | 9
Not completed — Adverse Event | 0 | 2 | 5 | 5 | 2 | 6
Not completed — Lack of Efficacy | 2 | 3 | 4 | 2 | 1 | 1
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other than specified above | 2 | 1 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sarilumab 100 mg q2w: Sarilumab 100 mg SC injection alternating with placebo q2w for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw | Total
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 50 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.7) | 42.4 (10.8) | 43.0 (11.3) | 40.4 (11.5) | 37.2 (10.4) | 41.1 (11.1) | 40.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 16 | 15 | 10 | 11 | 83
  Male | 38 | 30 | 34 | 37 | 40 | 39 | 218

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved 20% Response According to the Assessment in Ankylosing Spondylitis (AS) Working Group Criteria for Response (ASAS20) at Week 12
Description: Clinical response to treatment for ASAS20 was assessed according to ASAS20 criteria. Treatment response for ASAS20 was defined as an improvement by a decrease of ≥20% and ≥1unit on a 0 (no pain) - 10 (most severe pain) numerical rating scale (NRS) in at least 3 of the 4 ASAS improvement criteria (ASAS-IC) domains: assessment of physical function (measured by Bath Ankylosing Spondylitis Functional Index [BASFI]), back pain (0-10 NRS), participant global assessment (0-10 NRS) and inflammation (measured as the mean of the last 2 Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] questions) and no worsening (increase in score) of ≥20% and ≥1 unit on a 0-10 NRS in the remaining 4th domain.
Time Frame: Baseline to Week 12 (Last Observation Carried Forward [LOCF])
Population: Intent-to-treat (ITT) population included all randomized participants. Missing data was imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 50
percentage of participants | 24.0 | 24.5 | 30.0 | 19.2 | 30.0 | 38.0
Statistical Analysis 1: Comparison: Placebo vs Sarilumab 100 mg q2w; Sarilumab group was compared to placebo group. Analysis was performed using two-sided Cochran-Mantel-Haenszel test. Pairwise comparisons of the response rates between each dose of sarilumab and placebo were derived; Test type: Superiority or Other; p = 0.966, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.5]
Statistical Analysis 2: Comparison: Placebo vs Sarilumab 150 mg q2w; Test type: Superiority or Other; p = 0.467, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.6 to 3.5]
Statistical Analysis 3: Comparison: Placebo vs Sarilumab 100 mg qw; Test type: Superiority or Other; p = 0.559, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 1.9]
Statistical Analysis 4: Comparison: Placebo vs Sarilumab 200 mg q2w; Test type: Superiority or Other; p = 0.496, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.6 to 3.4]
Statistical Analysis 5: Comparison: Placebo vs Sarilumab 150 mg qw; Test type: Superiority or Other; p = 0.143, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.8 to 4.2]

2. Secondary Outcome: Percentage of Participants Who Achieved 40% Response According to the Assessment in AS Working Group Criteria for Response (ASAS40) at Week 12
Description: Clinical response to treatment for ASAS40 was assessed according to ASAS40 criteria. Treatment response for ASAS40 was defined as an improvement by a decrease of ≥40% and ≥2 units on a 0 (no pain)-10 (most severe pain) NRS in at least 3 of the 4 ASAS-IC domains (participant global assessment, back pain, physical function and inflammation) and no worsening (increase in score) at all in the remaining 4th domain.
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 50
percentage of participants | 8.0 | 14.3 | 16.0 | 5.8 | 18.0 | 20.0

3. Secondary Outcome: Percentage of Participants Who Achieved Partial Remission According to the Assessment in AS Working Group Criteria for Response (ASAS) at Week 12
Description: Participants were classified as having achieved ASAS partial remission if they had a value ≤ 2 units on a 0 -10 NRS in each of the 4 domains: (participant global assessment, back pain, physical function and inflammation) of the ASAS-IC.
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 50
percentage of participants | 2.0 | 8.2 | 2.0 | 1.9 | 2.0 | 8.0

4. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 12
Description: ASDAS consists of five components: (Total back pain assessed by BASDAI question 2 on a 0 [no pain] - 10 [most severe pain] NRS, participant global of disease activity on a 0 [none] - 10 [severe] NRS, peripheral pain/swelling assessed by BASDAI question 3 on a 0 [none] - 10 [most severe pain] NRS, duration of morning stiffness assessed by BASDAI question 6 on a NRS from 0 [0 hour] - 10 [2 or more hours] and hs-CRP in mg/L). ASDAS score was calculated as follows: 0.121 x total back pain + 0.110 x participant global of disease activity + 0.073 x peripheral pain/swelling + 0.058 x duration of morning stiffness + 0.579 x ln(CRP + 1). The scores were categorized as: inactive disease (< 1.3), moderate (1.3 - < 2.1), high (2.1 - 3.5) and very high disease activity (> 3.5).
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with ASDAS score assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 49 | 47 | 50 | 51 | 50 | 49
units on a scale | -0.4 (0.7) | -0.5 (0.9) | -0.8 (1.2) | -1.1 (0.8) | -1.2 (0.9) | -1.6 (0.9)

5. Secondary Outcome: Change From Baseline in BASDAI Score at Week 12
Description: BASDAI comprises of a 0 (no pain) -10 (very severe pain) NRS, used to answer 6 questions (Q) related to symptoms of AS (fatigue/tiredness, neck, back or hip pain, pain / swelling in joints, discomfort in tender areas, morning stiffness duration and morning stiffness severity). The BASDAI total score was calculated by computing the mean of Q5 and Q6 and adding it to the sum of Q1 to Q4. This score was then divided by 5. BASDAI total score=Q1+Q2+Q3+Q4+[Q5+Q6/2]/5. The total BASDAI score ranges from 0=none to 10=severe, where lower score indicated less disease activity.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with BASDAI score assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 50 | 49
units on a scale | -0.9 (1.7) | -0.8 (1.9) | -1.1 (2.0) | -0.4 (1.4) | -0.9 (1.8) | -1.2 (1.8)

6. Secondary Outcome: Change From Baseline in Range of Motion Assessed by the Bath AS Metrology Index (BASMI) at Week 12
Description: The range of motion was measured by the BASMI (11-point scale) including chest expansion in cm. It composed of 5 clinical measurements associated with a score: tragus to wall distance, modified schober's test, lateral spinal flexion, intermalleolar distance and cervical rotation. BASMI score was calculated by dividing the total of the score by 5, and the score ranges from 0-10. Higher BASMI score indicates more severe limitation of movement.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed=participants with BASMI score assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 50 | 49
units on a scale | -0.2 (0.8) | -0.2 (0.9) | -0.2 (0.8) | -0.4 (0.9) | -0.1 (0.8) | -0.2 (0.7)

7. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) Score of the Spine Assessed by the Berlin Modification of the AS Spine MRI-active (ASspiMRI-a) Score at Week 12
Description: ASspiMRI-a scoring system was used on all MRIs to score the level of the disease. MRIs were obtained using 1.0 or 1.5 Tesla scanners and phased array coils. Sagittal images of the upper (C2 to T10) and lower (T8 to S1) spine were used using both T1 weighted spin echo and fat saturated Short Tau Inversion Recovery (STIR) sequences. Each vertebral body unit was given an activity score based on the amount of bone marrow edema or erosion. Both T1 and STIR sequences were analyzed for change. Total spine ASspiMRI-a score in the Berlin modification range from 0 to 69 with higher scores indicating higher disease activity. A negative value in total spine ASspiMRI-a score change from baseline indicates an improvement from baseline. The higher the negative value the higher the reduction of inflammation.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = participants with ASspiMRI-a assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 45 | 42 | 44 | 47 | 46 | 44
units on a scale | -0.5 (2.2) | -0.5 (1.8) | -0.1 (3.4) | 0.1 (2.4) | -0.3 (3.3) | 0.3 (3.3)

8. Secondary Outcome: Percentage of Participants Who Achieved ASAS 5/6 Improvement Criteria at Week 12
Description: ASAS 5/6 responder had an improvement of 20% in 5 of 6 domains (physical function, back pain, participant global assessment, inflammation, spinal mobility and acute phase reactants) of ASAS-IC without deterioration in the 6th domain. Spinal mobility was assessed by the mean of the 5 BASMI scores on the 11-point scale (score ranges from 0-10) and the hs-CRP for the acute phase reactant.
Time Frame: Baseline to Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 50
percentage of participants | 6.0 | 12.2 | 10.0 | 13.5 | 14.0 | 32.0

9. Secondary Outcome: Change From Baseline in Chest Expansion at Week 12
Description: The difference between maximal inspiration and expiration to the nearest 0.1 cm was recorded. The best of 2 tries were recorded.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with chest expansion assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 49 | 47 | 49 | 51 | 50 | 49
cm | 0.2 (1.0) | 0.2 (1.2) | 0.0 (1.2) | -0.1 (0.9) | 0.1 (1.3) | 0.3 (1.3)

10. Secondary Outcome: Change From Baseline in Swollen Joint Index at Week 12
Description: 44 swollen joints were examined including sternal, clavicular, elbow, shoulder, wrist, knee, metacarpophalangian, interphalangian, metatarpophalangian and metatarsophalangeal joints.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with swollen joint count assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 48 | 50 | 51 | 50 | 49
Joints | -0.4 (1.1) | -0.8 (3.1) | -0.3 (1.9) | -0.3 (2.4) | -0.4 (1.6) | -0.2 (7.3)

11. Secondary Outcome: Change From Baseline in Hs-CRP at Week 12
Description: Participant's blood samples were collected at screening, baseline before dosing and at every visit to evaluate the level of hs-CRP. The hs-CRP is a protein marker in the blood associated with inflammation with higher values indicating a greater degree of inflammation.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with Hs-CRP assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Sarilumab 100 mg q2w | Sarilumab 150 mg q2w | Sarilumab 100 mg qw | Sarilumab 200 mg q2w | Sarilumab 150 mg qw
Number analyzed (Participants) | 50 | 48 | 50 | 51 | 50 | 49
mg/dL | -3.7 (19.1) | -1.2 (17.9) | -5.8 (27.6) | -13.5 (20.3) | -11.5 (17.5) | -14.3 (15.3)

12. Secondary Outcome: Change From Baseline in ASAS Individual Components at Week 12
Description: ASAS consists of 4 individual components: Participant global assessment to assess the disease activity over the last week on a 0 (no pain) - 10 (severe pain) NRS; back pain which consist of the mean of the nocturnal back pain and the total back pain at every visit on a 0 (no pain) - 10 (most severe pain) NRS; inflammation measured as the mean of the last 2 BASDAI questions (intensity and duration of morning stiffness) and physical function measured as mean of 10 scores of BASFI at every visit on 0 (easy) -10 (impossible) NRS. Lower score corresponds to a better functioning.
Time Frame: Baseline, Week 12 (LOCF)
Population: ITT population. Missing data was imputed using LOCF. Number of participants analyzed = participants with ASAS assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sarilumab 100mg q2w: Sarilumab 100 mg SC injection alternating with placebo q2w for 12 weeks.
- Sarilumab 150mg q2w: Sarilumab 150 mg SC injection alternating with placebo q2w for 12 weeks.
- Sarilumab 100mg qw: Sarilumab 100 mg SC injection qw for 12 weeks.
- Sarilumab 200mg q2w: Sarilumab 200 mg SC injection alternating with placebo q2w for 12 weeks.
- Sarilumab 150mg qw: Sarilumab 150 mg SC injection qw for 12 weeks.
Arm/Group | Placebo | Sarilumab 100mg q2w | Sarilumab 150mg q2w | Sarilumab 100mg qw | Sarilumab 200mg q2w | Sarilumab 150mg qw
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 50 | 49
units on a scale
  Participant global assessment | -1.0 (1.9) | -1.1 (2.3) | -0.8 (2.3) | -0.4 (2.2) | -0.9 (2.2) | -1.6 (2.0)
  Back pain | -0.8 (1.8) | -1.3 (2.2) | -1.2 (2.4) | -0.5 (1.8) | -0.9 (2.2) | -1.6 (2.1)
  Inflammation | -1.4 (1.8) | -0.8 (2.0) | -1.1 (2.0) | -0.7 (2.1) | -1.0 (1.9) | -1.8 (2.3)
  Physical function | -0.6 (1.2) | -0.5 (1.7) | -0.4 (2.0) | -0.1 (1.4) | -0.6 (1.9) | -1.1 (1.9)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 18) regardless of seriousness or relationship to investigational product
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during 'on treatment period' (time from first dose injection of double-blind study to end of 6-week follow-up period). Safety population included all randomized participants who received at least one dose of the study medication.
Groups:
- SAR153191 100 mg q2w: Sarilumab 100 mg SC injection alternating with placebo q2w for 12 weeks.
- SAR153191 150 mg q2w: Sarilumab 150 mg SC injection alternating with placebo q2w for 12 weeks. Included a participant randomized to sarilumab 200 mg q2w who received sarilumab 150 mg q2w in error.
- SAR153191 100 mg qw: Sarilumab 100 mg SC injection qw for 12 weeks.
- SAR153191 200 mg q2w: Sarilumab 200 mg SC injection alternating with placebo q2w for 12 weeks. Excluded a participant randomized to sarilumab 200 mg q2w who received sarilumab 150 mg q2w in error.
- SAR153191 150 mg qw: Sarilumab 150 mg SC injection qw for 12 weeks.
Arm/Group | Placebo | SAR153191 100 mg q2w | SAR153191 150 mg q2w | SAR153191 100 mg qw | SAR153191 200 mg q2w | SAR153191 150 mg qw
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/49 | 4/51 | 1/52 | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 7/50 | 18/49 | 23/51 | 22/52 | 19/49 | 22/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | SAR153191 100 mg q2w (N=49) | SAR153191 150 mg q2w (N=51) | SAR153191 100 mg qw (N=52) | SAR153191 200 mg q2w (N=49) | SAR153191 150 mg qw (N=49)
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
False positive tuberculosis test (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=50) | SAR153191 100 mg q2w (N=49) | SAR153191 150 mg q2w (N=51) | SAR153191 100 mg qw (N=52) | SAR153191 200 mg q2w (N=49) | SAR153191 150 mg qw (N=49)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 1 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 2 | 7 | 3 | 4
Viral infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 2 | 4 | 8
Headache (Nervous system disorders) | 0 | 4 | 2 | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 3 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 3 | 3 | 2 | 3 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 5 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 1
Fatigue (General disorders) | 0 | 3 | 2 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 3 | 1 | 1
Injection site pruritus (General disorders) | 0 | 0 | 1 | 3 | 0 | 1
Injection site reaction (General disorders) | 0 | 3 | 2 | 2 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 4 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 2 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.